CLINICAL TRIAL: NCT02479945
Title: Peripheral vs. Selective Tumor Marker Venous Sampling in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 06811
Record Dates: First submitted 2015-06-22; First posted 2015-06-24 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Selective internal iliac vein sampling (Other)
  Interventions: Other: Obtaining biospecimen

INTERVENTIONS:
Other: Obtaining biospecimen

SUMMARY:
The investigators will compare tumor marker levels, including PSA, in samples taken from a peripheral upper limb vein and the internal iliac veins. These will be collected from patients who are scheduled for prostatectomy as part of their standard of care for prostate cancer. A selective internal iliac vein sampling procedure will be performed in Interventional Radiology. Venous samples will be correlated with prostatectomy specimens. The aim is to predict the side of the prostate containing tumor.

ELIGIBILITY:
Inclusion Criteria:

1. All male patients, age 18 to 99, with biopsy proven prostate adenocarcinoma prior to planned radical prostatectomy.
2. Informed Consent/HIPAA Form discussed and signed by subject.
3. Baseline lab values obtained within 120 days of planned selective venous sampling.

Exclusion Criteria:

1. Skin related problems around the planned venepuncture site (infection, phlebitis, scars)
2. Documented allergy to iodinated contrast or lidocaine.
3. Coagulopathy with an INR of greater than 1.5
4. Thrombocytopenia with platelets less than 25,000 uL
5. Renal insufficiency with a creatinine of 1.5 mg/dL
6. Documented current upper extremity or central venous thrombosis
7. DRE within 4 weeks prior to selective venous sampling
8. Prostate biopsy within 6 weeks prior to selective venous sampling.
9. Patient unable to sign his own consent or does not demonstrate full understanding of the procedure.
10. Patient has known metastatic disease or a known primary cancer other than prostate adenocarcinoma.
11. Patient has already been enrolled in this research study.
12. Life expectancy less than 6 months.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-04-25 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Micah Watts, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States